CLINICAL TRIAL: NCT00681668
Title: The Effect of the Atypical Antipsychotic Quetiapine in the Treatment of Postpartum Depressive Disorder With Psychotic Symptoms
Brief Title: Quetiapine in Postpartum Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment behind plan, no increase expected
Sponsor: AstraZeneca (Industry)
Responsible Party: Kai Richter MD, Medical Director (comm), MC Germany, AstraZeneca, MC Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1449L00023
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Postpartum Depressive Disorder
Keywords: Postpartum Depression; Quetiapine; Psychotic Symptoms
MeSH Terms: conditions — Depression, Postpartum | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine Fumarate 150 - 800mg (Experimental): Quetiapine 150-800mg
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — 150-800 mg, oral, twice a day (bid)
  Other Names: Seroquel

SUMMARY:
The purpose of the study is to evaluate the efficacy and tolerability of quetiapine in female patients with postpartum depressive disorder with psychotic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent.
* Female patients with severe postpartum depressive disorders with psychotic symptoms and a minimum HAM-D cut off score of 20 points

Exclusion Criteria:

* Woman with pre-existing psychotic disorder
* Patients with alcohol or substance abuse or dependence
* Patients who pose an imminent risk of suicide or danger to self or others

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Turmes, MD, Principal Investigator — Westfälisches Zentrum Herten, Psychiatrie und Psychotherapie Im Schlosspark 20 45699 Herten
Locations (1):
- Research Site, Herten, Westfalen-Lippe, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period July 2007 to October 2008; Medical Clinic - Westfälischen Zentrums Herten; Psychiatrie and Psychotherapie
Groups:
- Quetiapine Fumarate 150 - 800mg: Quetiapine fumarate, tablets, 150 - 800mg oral, per day, until 28 weeks
Period: Overall Study
Arm/Group | Quetiapine Fumarate 150 - 800mg
Started | 5
Completed | 3
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine Fumarate 150 - 800mg
Number analyzed (Participants) | 5
Age, Customized [Number; unit: Participants]
  18 to < 40 years | 5
  Between 18 and 65 years | 0
  >= 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Hamilton Rating Scale for Depression (HAM-D)
Description: HAM-D is a 17-21 item observer-rated scale to assess presence and severity of depressive states. 9 items are scored 0-4, whereas the further 8 are scored 0-2, as these represent variables which do not lend themselves to quantitative rating (0=absent; 1=doubtful or slislight; 2=clearly present). Higher scores indicate higer depressive state
Time Frame: Baseline Day 1 to final visit 28 weeks
Measure: Mean (Full Range); unit: scores on a HAM-D scale
Groups:
- Quetiapine Fumarate: Quetiapine fumarate tablets
Arm/Group | Quetiapine Fumarate
Number analyzed (Participants) | 5
scores on a HAM-D scale | 21 [7 to 26]

2. Secondary Outcome: Change in Efficacy Scales: Clinical Global Impression (CGI), Montgomery Asberg Depression Rating Scale (MADRS), Brief Psychiatric Rating Scale (BPRS)
Description: Change in efficacy scales: Clinical Global Impression (CGI),Scale of 1-7 (1 = normal or no change - 7 = extremely ill or extreme changes).
  Montgomery Asberg Depression Rating scale (MADRS) 10 questions with a scale of 1-4 (1 = no symptoms - 4 = severe symptoms), higher score = worst values.
  Brief Psychiatric rating scale (BPRS)- 24 symptom constructs, each to be rated in a 7-point scale of severity ranging from 'not present' to 'extremely severe' no participants analysed - terminated study
Time Frame: Baseline Day 1 to final visit 28 weeks
Population: Data not analyzed, study terminated
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Quetiapine Fumarate
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Functional Outcome: Global Assessment of Functioning (GAF), Parental Bonding Questionnaire (PBQ)
Description: Change in functional outcome: Global Assessment of Functioning (GAF),scale of 1-100 (1 = severe symptoms - 100 = no symptoms) Parental bonding Questionnaire (PBQ) no participants analysed - terminated study
Time Frame: Baseline Day 1 to final visit 28 weeks
Population: Data not analyzed, study terminated
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Quetiapine Fumarate
Number analyzed (Participants) | 0

4. Secondary Outcome: Electrocardiogram (ECG), Vital Signs, Laboratory
Description: Safety parameter:s electrocardiogram (ECG), vital signs, laboratory
  no participants analysed - terminated study
Time Frame: Baseline Day 1 to final visit 28 weeks
Population: Data not analyzed, study terminated
Measure: Number; unit: participants
Arm/Group | Quetiapine Fumarate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Quetiapine Fumarate 150 - 800mg
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Quetiapine Fumarate 150 - 800mg
Nasopharyngitis (Infections and infestations) | 2/5
Diarrhoea (Gastrointestinal disorders) | 1/5
Eczema (Skin and subcutaneous tissue disorders) | 1/5
Gastritis (Gastrointestinal disorders) | 1/5

LIMITATIONS AND CAVEATS:
Study termination (the study could not finalised in the planned,nor in an acceptable time).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site has to inform sponsor about a publication at least 60 day in advance and 10 days before submission of an abstract or presenation. Change requests by the sponsor are recognized unless the scientific character or the objectivity is on risk. If the sponsor plans a patent applicaion the publication has to be postponed up to 120 days.